CLINICAL TRIAL: NCT02568527
Title: Study to Evaluate Safety & Efficacy of PLGA Scaffold to Regenerate Limbal Epithelial Cells Using Autologous Limbal Grafts by SLET (Simple Limbal Epithelial Transplant) Procedure in Patients Having Total Unilateral LSCD
Brief Title: Biodegradable Synthetic Scaffold as a Substitute for hAM in Limbal Epithelial Cells Transplant in LSCD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virender S Sangwan, MBBS, MS (Other)
Collaborators: Wellcome Trust (Other); University of Sheffield (Other)
Responsible Party: Sponsor-Investigator, Virender S Sangwan, MBBS, MS, Director, Center for Ocular Regeneration (CORE), L.V. Prasad Eye Institute
Organization: L.V. Prasad Eye Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LVPEI-2012-11
Record Dates: First submitted 2015-08-27; First posted 2015-10-06 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2016-04

CONDITIONS: Limbal Stem Cell Deficiency
Keywords: LSCD; SLET; Donor Human Amniotic Membrane (hAM); PLGA
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PLGA Scaffold (Experimental): Poly Lactide-co-Glycolic Acid (PLGA) 50:50
  Interventions: Device: PLGA scaffold

INTERVENTIONS:
Device: PLGA scaffold — Poly-Lactic-co-Glycolic Acid (50:50) biodegradable, synthetic scaffold
  Other Names: Purasorb PDLG 5004

SUMMARY:
The purpose of this clinical study is to undertake a pilot safety and efficacy study of a synthetic biodegradable membrane as a substitute for using donor human amniotic membrane (hAM) for the treatment of limbal stem cell deficiency (LSCD) by combining this with freshly excised limbal tissue in theatre as a one stage procedure

DETAILED DESCRIPTION:
This study will involve the used of a synthetic biodegradable Poly Lactide-co-Glycolic Acid (PLGA) biodegradable, synthetic carrier membrane (PLGA) membrane as a substitute for using donor human amniotic membrane (hAM) for the treatment of limbal stem cell deficiency (LSCD) by combining this with freshly excised limbal tissue in theatre as a one stage procedure.

This has the potential to simplify the current procedure and make it safer and accessible to more surgeons and eventually benefit more patients. The use of PLGA membrane, in place of hAM for limbal transplants, is a novel technique and has a lot of promise and potential, which will potentially benefit patients at large and significantly bring down costs for the limbal transplants while reducing the disease transmission risks of using human donor tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants who are ≥18 years of age.
2. Patients having a confirmed diagnosis of total LSCD as confirmed by any one or all of the following:

   * In-growth of conjunctival epithelium over the cornea (conjunctivalization),
   * 360o absence of limbal Palisades of Vogt,
   * A fine stippled appearance on fluorescein staining,
   * Persistent or recurrent corneal epithelial defects
   * Superficial vascularization,
   * Dull and irregular corneal epithelium.
3. Participants having unilateral limbal stem cell deficiency due to chemical injury
4. No prior history of limbal transplantation
5. No ongoing and other active ocular pathology
6. No severe pathological and psychological conditions that might interfere with the patients participation in the study
7. Able to provide written informed consent prior to any study specific screening procedures with the understanding that the patient has the right to withdraw from the study at any time, for any reason without prejudice.

Exclusion Criteria:

1. Bilateral LSCD
2. LSCD due to autoimmune disorders and partial LSCD
3. Having other ongoing ocular pathologies and acute ocular inflammation
4. Previous neoplastic/cancer disease
5. Severe dry eyes confirmed by Schirmer's test
6. Acute systemic infections
7. Prior history of limbal transplantation surgery or multiple surgeries in the limbal region
8. Substance abuse, medical, psychological or social conditions that may, in the opinion of the investigator, interfere with the patient's participation in the study or evaluation of the study results.
9. Any uncontrolled, inter-current illness that in the opinion of the Investigator may interfere with study evaluation.
10. Participants with uncontrolled diabetes will be excluded from the study
11. History or evidence of cardiac disease: congestive heart failure; New York Heart Association (NYHA) class 2 or greater (see Appendix 6); active coronary artery disease; unstable angina, cardiac arrhythmias requiring anti-arrhythmic therapy, atrio-ventricular block of second or third degree, or uncontrolled hypertension, patients with recent (less than 6 months) myocardial infarction (MI) or coronary revascularization.
12. Pregnant and lactating patients, positive urine pregnancy test in women of childbearing potential
13. Reproductive age patients not practicing effective and adequate birth control measures
14. Participation in any other investigational trial in which receipt of investigational drug or device occurred within 30 days prior to screening for this study.
15. Previous participation in this study

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Corneal Edema using Pachymetry | 12 months
  At Baseline and at Month 12
Intraocular Pressure by Standard Applanation Tonometry | 12 months
  At Baseline and at Month 12
Ocular Pain | 12 months
  Magnitude of pain will assessed as patient reported outcome using Visual Analogue Scale (VAS) in a scale of 1 to 10 (Wong-Baker Faces Pain Rating Scale)
Schirmer's test (5 minute) without anesthesia | 12 months
Clinical Laboratory Adverse Events | 12 months
Vital Signs | 12 months

SECONDARY OUTCOMES:
Regeneration of Stable Ocular Surface measured by Slit lamp Biomicroscopy Examination and Slit Lamp Photography | 12 months
Best Corrected Visual Acuity by Snellen Chart | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Virender S Sangwan, MBBS MS, Principal Investigator — LV Prasad Eye Institute; Sayan Basu, MBBS MS, Study Director — LV Prasad Eye Institute
Locations (1):
- LV Prasad Eye Institute, Hyderabad, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: No